CLINICAL TRIAL: NCT04601701
Title: Study on Central Retinal Vein Occlusion Patients Receiving Bevacizumab and Dexamethasone or Bevacizumab Only on Naive Eyes.
Brief Title: Central Retinal Vein Occlusion (CRVO) Treatment With Bevacizumab and Dexamethasone or Bevacizumab Only.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ME-270620
Record Dates: First submitted 2020-08-26; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Bevacizumab; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRVO: Bevacizumab and intravitreal Dexamethasone. (Experimental): Participants with CRVO will receive a combination of Bevacizumab and intravitreal Dexamethasone.
  Interventions: Drug: Bevacizumab Ophthalmic and Intravitreal Dexamethasone.
- CRVO: Bevacizumab (Active Comparator): Participants with CRVO will receive a combination of Bevacizumab only.
  Interventions: Drug: Bevacizumab Ophthalmic.

INTERVENTIONS:
Drug: Bevacizumab Ophthalmic and Intravitreal Dexamethasone. — Pro re nata patients with CRVO will initially receive Bevacizumab and intravitreal Dexamethasone. And then depending on their clinical status of CRVO, Bevacizumab will be injected.
  Other Names: Avastin®; Ozurdex®
  Arms: CRVO: Bevacizumab and intravitreal Dexamethasone.
Drug: Bevacizumab Ophthalmic. — Pro re nata patients with CRVO will receive Bevacizumab. And then depending on their clinical status of CRVO, Bevacizumab will be injected.
  Other Names: Avastin®
  Arms: CRVO: Bevacizumab

SUMMARY:
The purpose of this study is to determine whether Bevacizumab (Avastin) in combination with Dexamethasone (Ozurdex) will be effective in reducing if not eliminating the macular edema associated with the disease, central retinal vein occlusion (CRVO) in comparison to Bevacizumab (Avastin) alone.

DETAILED DESCRIPTION:
Retinal Venous Occlusive disease is the second only to diabetic retinopathy as a major cause of blindness associated with retinal vascular disease. Macular edema is a major cause of vision loss in patients presenting with central and hemi vein occlusions. Until recently the standard of care for macular edema secondary to central retinal vein occlusion was observation. Recent investigations of steroids for this condition has shown greater visual benefit but is associated with risks such as cataract formation and increased intraocular pressure. In the past laser photocoagulation has been used, but was found to offer no visual benefits over the natural history in the treatment of macular edema associated with CRVO.

Bevacizumab, an anti-VEGF agent, is a potent inhibitor of vascular permeability, with the potential to reduce retinal vascular leakage and diminish macular edema. In addition, as an anti-VEGF agent, it may also inhibit neovascularization of the iris, a frequent complication of ischemic central retinal vein occlusion. Bevacizumab use as an intravitreal agent does carry the risk of intraocular infection but probably carries very low risk of glaucoma or cataract formation, making it a potentially safer pharmacologic treatment for CRVO associated macular edema as compared to steroids.

Ozurdex (dexamethasone) Intravitreal Implant is a steroid injected into the eye to treat swelling that may occur when there is a blockage of certain blood vessels in your eyes. Ozurdex is also used to treat non-infectious uveitis affecting the posterior (rear) segment of the eye.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any study assessment is performed
2. Diagnosis of visual impairment exclusively due to ME secondary to CRVO
3. BCVA score at Screening and Baseline between 73 and 19 letters (ETDRS)

Exclusion Criteria:

1. Pregnant or nursing (lactating) women
2. Stroke or myocardial infarction less than 3 months before Screening
3. Uncontrolled blood pressure defined as systolic value of >160 mm Hg or diastolic value of >100 mm Hg at Screening or Baseline.
4. Any active periocular or ocular infection or inflammation at Screening or Baseline in either eye
5. Uncontrolled glaucoma at Screening or Baseline or diagnosed within 6 months before Baseline in either eye
6. Neovascularization of the iris or neovascular glaucoma in the study eye
7. Use of any systemic antivascular endothelial growth factor (anti-VEGF) drugs within 6 months before Baseline
8. Panretinal laser photocoagulation within 3 months before Baseline or anticipated or scheduled within the next 3 months following Baseline in the study eye
9. Focal or grid laser photocoagulation within 4 months before Baseline in the study eye
10. Use of intra- or periocular corticosteroids (including sub-Tenon) or ocular anti-VEGF treatment within 3 months before Screening in the study eye
11. Any use of intraocular corticosteroid implants (eg, dexamethasone [Ozurdex®], fluocinolone acetonide [Iluvien®]) in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-09-17 (Estimated)

PRIMARY OUTCOMES:
Mean change in monocular BCVA in the treatment eye | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Monocular BCVA in the treatment eye is assessed by using ETDRS visual acuity charts at 4 meters.
Mean change in binocular BCVA | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Binocular BCVA is assessed by using ETDRS visual acuity charts at 4 meters.

SECONDARY OUTCOMES:
Mean change in central subfield retinal thickness | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean change in central subfield retinal thickness in the study eye, as determined by spectral domain optical coherence tomography (OCT).
Change in Humphrey 10-2 visual field in the treatment eye | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of the Humphrey 10-2 visual field is assessed by a Humphrey 10-2 visual field test.
Number of Ranibizumab Treatments | Day 1 through Month 6
  Number of injections provided to the patients during the 6 month period.
Mean change in NEI VFQ25 Questionnaire Score | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Scores from NEI VFQ25 questionnaire will be assessed and compared
Mean change in VisQoL scores | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Scores from VisQoL questionnaire will be assessed and compared
Mean change in wavefront aberrations | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of wavefront aberrations is assessed by Nidek OPD Scan III test
Mean change in ocular surface and tear-film | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of ocular surface and tear-film parameters is assessed by Oculus Keratographer test
Mean change in vessel density | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Mean deviation (MD) of vessel density is assessed by Spectralis OCT2, Heidelberg-Engineering test
Side effects | Baseline, 1 week, 1 month, 2 months, 3 months, and 6 months.
  Side effects are measured by a review of the participant's medical and ophthalmic history.
Use of additional treatments (including laser) | Day 1 through Month 6
  Use of additional treatments (including laser) is assessed by the treating ophthalmologist
People meeting driving standards | Baseline, 1 week, 1month, 2 months, 3 months, and 6 months.
  Percentage (%) of people meeting driving standards is assessed by an Esterman binocular visual field test

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, M.D., Ph.D., Study Chair — He Eye Specialist Hospital, Shenyang.; Jun Li, M.D., Ph.D., Principal Investigator — He Eye Specialist Hospital, Shenyang.; Emmanuel E Pazo, M.D., Ph.D., Study Director — He Eye Specialist Hospital, Shenyang.
Locations (1):
- He Eye Specialist Hospital, Shenyang, Liaoning, China